CLINICAL TRIAL: NCT04292951
Title: Early Goal Directed Therapy vs Standard Protocol for Hemodynamic Management in Patients Undergoing Cardiac Surgery: A Randomized Controlled Trial
Brief Title: Early Goal Directed Therapy in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE611321
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Outcome; ICU Stay
Keywords: Postoperative outcome; Goal directed therapy; Arterial pressure derived cardiac output
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Group GDT: fluid and inotropic/vasoactive drugs management guided by FloTrac/EV1000 Group Control: fluid and inotropic/vasoactive drugs management guided by central venous pressure (CVP), blood pressure, heart rate, and clinical signs
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient is anesthetized, thus unaware type of treatment. The assessor is blinded of the monitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDT group (Experimental): Intraoperative fluid and inotropic/vasoactive drugs management based on information from FloTrac/EV1000
  Interventions: Procedure: Fluid and inotropic/vasoactive management protocol
- Control group (Active Comparator): Intraoperative fluid and inotropic/vasoactive drugs management based on CVP, blood pressure, heart rate, and clinical signs at the discretion of attending anesthesiologists
  Interventions: Procedure: Fluid and inotropic/vasoactive management protocol

INTERVENTIONS:
Procedure: Fluid and inotropic/vasoactive management protocol — GDT protocol: keep SVV 10-13% and give fluid when SVV > 13%, give inotropic to maintain CI 2.5-4 L/min/m2, give vasoactive drugs to maintain SVRI 1,900-2,400 dynes-sec/cm-5/m2 Control protocol: keep CVP 8-12 mmHG and give fluid when CVP < 8 mmHg, give inotropic/vasoactive to maintain normal blood pressure and heart rate

SUMMARY:
Early goal directed therapy (EGDT) based on information from arterial waveform derived cardiac output (APCO) FloTrac/EV1000 system has been proved to improve postoperative outcomes in patients undergoing major surgery. This system, however, has the limitation to be applied in open-chest surgery, especially cardiac surgery. The efficiency of FloTrac/EV1000 system to improve postoperative outcomes in cardiac surgery is still inconclusive.

Hypothesis: Intraoperative management in patients undergoing cardiac surgery guided by FloTrac/EV1000 system, compared with conventional protocol, results in better clinical outcomes.

Primary outcomes: Immediate postoperative inotropic/vasoactive drugs requirement.

Methods: Adult patients undergoing cardiac surgery will be randomized into 2 groups: EGDT group managed by FloTrac/EV1000 system and Control group managed by conventional protocol.

Outcome analyses: Compare the number of inotropic/vasoactive drugs requirement at the end of surgery, as well as intensive care unit (ICU) stay between both groups.

DETAILED DESCRIPTION:
Objective: To compare postoperative clinical outcome in adult patients undergoing cardiac surgery.

Primary outcome: Postoperative inotropic/vasoactive drugs reqirement.

Secondary outcome: ICU stay.

Methods: Eligible patients will be randomized to 2 groups. Both groups will be managed intraoperatively in the same way, except fluid and inotropic/vasoactive drugs management protocol. EGDT group will be managed according to information derived from FloTrac/EV1000 system, i.e., control stroke volume variation (SVV) 10-13% and give fluid when SVV > 13%, give inotropic to maintain cardiac index (CI) 2.5-4 L/min/m2, and give vasoactive drugs to maintain systemic vascular resistance index (SVRI) of 1,900-2,400 dynes-sec/cm-5/m2 . Control group will be managed using central venous pressure (CVP) protocol, i.e., control CVP 8-12 mmHg and give fluid when CVP < 8 mmHg, give inotropic/vasoactive drugs according to blood pressure and heart rate as well as clinical signs at the discretion of attending anesthesiologists.

Outcome analyses: Postoperative number of inotropic/vasoactive drugs requirement as well as ICU stay of both groups will be compared using unpaired Student-t test or Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Patient has ischemic or valvular heart disease
3. Scheduled for elective cardiac surgery
4. New York Heart Association (NYHA) or American society of Anesthesiology (ASA) classification I-III
5. Body mass index (BMI) 18-24 kg/m2
6. Provided informed consent before surgery

Exclusion Criteria:

1. Scheduled for emergency or redo surgery
2. Difficulty (or contraindication to) placing a central venous catheter
3. Inability to cooperate (e.g. mental disorder, disturbance of consciousness, mental retardation)
4. Presence of blood-borne infectious disease (e.g. syphilis, acquired immunodeficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Number of inotropic/vaso active drugs requirement | up to Day 1 postoperatively
  number of inotropic/vasoactive drugs required to maintain normal blood pressure and heart rate

SECONDARY OUTCOMES:
ICU stay | up to day 10 postoperatively
  number of hours admitted in ICU
Lactate level | up to Day 1 postoperatively
  serum lactate level
Creatinine level | up to day 10 postoperatively
  serum creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD, Study Chair — Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bednarczyk JM, Fridfinnson JA, Kumar A, Blanchard L, Rabbani R, Bell D, Funk D, Turgeon AF, Abou-Setta AM, Zarychanski R. Incorporating Dynamic Assessment of Fluid Responsiveness Into Goal-Directed Therapy: A Systematic Review and Meta-Analysis. Crit Care Med. 2017 Sep;45(9):1538-1545. doi: 10.1097/CCM.0000000000002554. PMID 28817481
- [Result] Kapoor PM, Kakani M, Chowdhury U, Choudhury M, Lakshmy, Kiran U. Early goal-directed therapy in moderate to high-risk cardiac surgery patients. Ann Card Anaesth. 2008 Jan-Jun;11(1):27-34. doi: 10.4103/0971-9784.38446. PMID 18182756
- [Result] Kusaka Y, Ohchi F, Minami T. Evaluation of the Fourth-Generation FloTrac/Vigileo System in Comparison With the Intermittent Bolus Thermodilution Method in Patients Undergoing Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):953-960. doi: 10.1053/j.jvca.2018.06.017. Epub 2018 Jun 28. PMID 30077561
- [Result] Lopes MR, Oliveira MA, Pereira VO, Lemos IP, Auler JO Jr, Michard F. Goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery: a pilot randomized controlled trial. Crit Care. 2007;11(5):R100. doi: 10.1186/cc6117. PMID 17822565
- [Derived] Tribuddharat S, Sathitkarnmanee T, Ngamsaengsirisup K, Sornpirom S. Efficacy of early goal-directed therapy using FloTrac/EV1000 to improve postoperative outcomes in patients undergoing off-pump coronary artery bypass surgery: a randomized controlled trial. J Cardiothorac Surg. 2022 Aug 21;17(1):196. doi: 10.1186/s13019-022-01933-4. PMID 35989328